CLINICAL TRIAL: NCT04145531
Title: An Open-Label, Multicenter Study of Recombinant Crisantaspase Produced in Pseudomonas Fluorescens (RC-P) in Patients With Acute Lymphoblastic Leukemia (ALL)/Lymphoblastic Lymphoma (LBL) Following Hypersensitivity to E. Coli-derived Asparaginases
Brief Title: An Open-Label Study of JZP-458 (RC-P) in Patients With Acute Lymphoblastic Leukemia (ALL)/Lymphoblastic Lymphoma (LBL)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JZP458-201; AALL1931 (Other: Children's Oncology Group)
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Acute Lymphoblastic Leukemia; Lymphoblastic Leukemia
Keywords: ALL; LBL; Asparaginase; Leukemia; Childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JZP-458 (Experimental): Part A (IM JZP-458) of the study will have 2 IM cohorts:
  * Cohort 1: a JZP-458 repeat dose/confirmatory cohort; a final IM JZP-458 dose level will be selected, and
  * Cohort 2: an expansion cohort to confirm the efficacy and safety of the final IM JZP-458 dose level and schedule
  Part B (IV JZP-458 Dose Confirmation) will be conducted to define the optimal dose of the IV administration of JZP-458 for further study in ALL/LBL patients as a repeated dose.
  Additional courses of JZP-458 (IM or IV depending on patient's allocation at study enrollment) will be administered based on each patient's original treatment plan for as long as the patient derives clinical benefit.
  Interventions: Drug: IM JZP-458; Drug: IV JZP-458

INTERVENTIONS:
Drug: IM JZP-458 — IM JZP-458 will be administered in Part A, Cohorts 1 & 2
Drug: IV JZP-458 — IV JZP-458 will be administered in Part B

SUMMARY:
This is an open-label, multicenter, dose confirmation, and PK study of JZP-458 in patients (of any age) with ALL/LBL who are hypersensitive to E. coli-derived asparaginases (allergic reaction or silent inactivation). This study is designed to assess the tolerability and efficacy of JZP-458 (only in patients who develop hypersensitivity to an E. coli-derived asparaginase), as measured by asparaginase activity.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric and adult patients with a diagnosis of ALL or LBL.
2. Have had an allergic reaction to a long-acting E. coli-derived asparaginase OR have silent inactivation.
3. Have 1 or more courses of E. coli-derived asparaginase remaining in his/her treatment plan.
4. Patients must have, in the opinion of the Investigator, fully recovered from their prior allergic reaction to E. coli-derived asparaginase.

Exclusion Criteria:

1. Have previously received asparaginase Erwinia chrysanthemi or JZP-458.
2. Have relapsed ALL or LBL.
3. Are concurrently receiving another investigational agent and/or treated with an investigational device at the same time as JZP-458 (within 48 hours) during Course 1 of JZP-458.
4. Have a history of ≥ Grade 3 pancreatitis.
5. Prior history of asparaginase-associated ≥ Grade 3 hemorrhagic event or asparaginase-associated thrombus requiring anticoagulation therapy, excluding catheter-related thrombotic events.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2019-12-27 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-07-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (74):
- United States (67):
  - Children's of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente - Orange County - Anaheim Medical Center, Anaheim, California
  - Kaiser Permanente - Downey Medical Center, Downey, California
  - Kaiser Permanente - Fontana Medical Center, Fontana, California
  - Loma Linda University Medical Center, Loma Linda, California
  - MemorialCare Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Kaiser Permanente- Los Angeles Medical Center, Los Angeles, California
  - Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente - Oakland Medical Center, Oakland, California
  - Children's Hospital of Orange County Main Campus - Orange, Orange, California
  - Kaiser Permanente - Roseville Medical Center, Roseville, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente - San Diego Medical Center, San Diego, California
  - University of California San Francisco Benioff Children's Hospital - Mission Bay, San Francisco, California
  - Kaiser Permanente - Santa Clara Medical Center, Santa Clara, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Smilow Cancer Hospital - New Haven, New Haven, Connecticut
  - Nemours Alfred I. Dupont Hospital for Children, Wilmington, Delaware
  - Children's National Health System, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Memorial Medical Office Centre, Hollywood, Florida
  - Nemours Children's Specialty Care Jacksonville, Jacksonville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Scottish Rite Hospital, Atlanta, Georgia
  - Kapi'olani Medical Center for Women and Children, Honolulu, Hawaii
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Norton Children's Hospital, Louisville, Kentucky
  - Dana-Farber/Boston Children's Cancer and Blood Disorders Center, Boston, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Minnesota, Minneapolis, Minnesota
  - Masonic Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University School of Medicine in Saint Louis, St Louis, Missouri
  - Alliance for Childhood Diseases, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Cohen Children's Medical Center, New Hyde Park, New York
  - NYU - Stephen D. Hassenfeld Children's Center for Cancer and Blood Disorders, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center - New York, New York, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Children's Hospital at Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Neurology Clinic, P.C, Cordova, Tennessee
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Children's Blood and Cancer Center, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Methodist Hospital - San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Inova Medical Group - Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center, Spokane, Washington
- Canada (7):
  - CancerCare Manitoba - McDermot and Urgent Care Site, Winnipeg, Manitoba
  - McMaster Children's Hospital, Hamilton, Ontario
  - Victoria Hospital & Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - SickKids - The Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - The Montreal Children's Hospital, Montreal, Quebec

REFERENCES:
- [Result] Maese L, Loh ML, Choi MR, Lin T, Aoki E, Zanette M, Agarwal S, Iannone R, Silverman JA, Silverman LB, Raetz EA, Rau RE. Recombinant Erwinia asparaginase (JZP458) in acute lymphoblastic leukemia: results from the phase 2/3 AALL1931 study. Blood. 2023 Feb 16;141(7):704-712. doi: 10.1182/blood.2022016923. PMID 36108304
- [Derived] Maese L, Loh ML, Choi MR, Agarwal S, Aoki E, Liang Y, Lin T, Girgis S, Chen C, Roller S, Chandrasekaran V, Iannone R, Silverman LB, Raetz EA, Rau RE. Recombinant Erwinia asparaginase (JZP458) in ALL/LBL: complete follow-up of the Children's Oncology Group AALL1931 study. Blood Adv. 2025 Jan 14;9(1):66-77. doi: 10.1182/bloodadvances.2024013346. PMID 39454281

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 229 participants who met all inclusion and no exclusion criteria were enrolled in the study. One participant did not receive treatment; 228 participants were included in the Safety Analysis Set and 224 participants were included in the Efficacy Analysis Set. The data presented are based on the final database cut (22 November 2022).
Groups:
- Part A: JZP-458 IM 25 mg/m^2 (MWF): Participants who received an intramuscular (IM) dose of JZP-458 25 mg/m^2 on a Monday/Wednesday/Friday (MWF) schedule over 2 weeks based on available data from the Phase 1 (JZP458-101) healthy volunteer study.
- Part A: JZP-458 IM 37.5 mg/m^2 (MWF): Participants who received an intramuscular (IM) dose of JZP-458 37.5 mg/m^2 on a Monday/Wednesday/Friday (MWF) schedule over 2 weeks.
- Part A: JZP-458 IM 25 (MW)/50 mg/m^2 (F): Participants who received an intramuscular (IM) dose of JZP-458 25 mg/m^2 on Mondays and Wednesdays and 50 mg/m^2 on Fridays on a Monday/Wednesday/Friday (MWF) schedule over 2 weeks.
- Part B: JZP-458 IV 25 (MW)/50 mg/m^2 (F): Participants who received an intravenous (IV) dose of JZP-458 25 mg/m^2 on Mondays and Wednesdays and 50 mg/m^2 on Fridays on a Monday/Wednesday/Friday (MWF) schedule over 2 weeks.
Period: Part A
Arm/Group | Part A: JZP-458 IM 25 mg/m^2 (MWF) | Part A: JZP-458 IM 37.5 mg/m^2 (MWF) | Part A: JZP-458 IM 25 (MW)/50 mg/m^2 (F) | Part B: JZP-458 IV 25 (MW)/50 mg/m^2 (F)
Started | 33 | 83 | 51 | 0
Safety Analysis Set | 33 | 83 | 51 | 0
Efficacy Analysis Set | 32 | 83 | 50 | 0
Completed | 27 | 62 | 39 | 0
Not Completed | 6 | 21 | 12 | 0
Not completed — Adverse Event | 2 | 12 | 6 | 0
Not completed — Death | 1 | 2 | 0 | 0
Not completed — Physician Decision | 2 | 5 | 2 | 0
Not completed — Progressive disease | 0 | 2 | 1 | 0
Not completed — Protocol deviation | 0 | 0 | 1 | 0
Not completed — Withdrawal by parent or guardian | 1 | 0 | 0 | 0
Not completed — Withdrawal by participant | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 1 | 0
Period: Part B
Arm/Group | Part A: JZP-458 IM 25 mg/m^2 (MWF) | Part A: JZP-458 IM 37.5 mg/m^2 (MWF) | Part A: JZP-458 IM 25 (MW)/50 mg/m^2 (F) | Part B: JZP-458 IV 25 (MW)/50 mg/m^2 (F)
Started | 0 | 0 | 0 | 62
Safety Analysis Set | 0 | 0 | 0 | 61
Efficacy Analysis Set | 0 | 0 | 0 | 59
Completed | 0 | 0 | 0 | 27
Not Completed | 0 | 0 | 0 | 35
Not completed — Adverse Event | 0 | 0 | 0 | 21
Not completed — Physician Decision | 0 | 0 | 0 | 7
Not completed — Progressive disease | 0 | 0 | 0 | 1
Not completed — Recurrent disease | 0 | 0 | 0 | 1
Not completed — Withdrawal by parent or guardian | 0 | 0 | 0 | 3
Not completed — Withdrawal by participant | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics were assessed in the Safety Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: JZP-458 IM 25 mg/m^2 (MWF) | Part A: JZP-458 IM 37.5 mg/m^2 (MWF) | Part A: JZP-458 IM 25 (MW)/50 mg/m^2 (F) | Part B: JZP-458 IV 25 (MW)/50 mg/m^2 (F) | Total
Number analyzed (Participants) | 33 | 83 | 51 | 61 | 228
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25 | 79 | 46 | 54 | 204
  Between 18 and 65 years | 8 | 4 | 5 | 7 | 24
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.5 (7.11) | 9.0 (5.08) | 11.3 (5.41) | 10.4 (6.30) | 10.3 (5.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 28 | 20 | 25 | 89
  Male | 17 | 55 | 31 | 36 | 139
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 3 | 2 | 5
  Asian | 1 | 5 | 1 | 3 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 11 | 8 | 2 | 24
  White | 24 | 58 | 33 | 43 | 158
  More than one race | 1 | 0 | 0 | 1 | 2
  Unknown or Not Reported | 4 | 9 | 6 | 10 | 29

OUTCOME MEASURES:

1. Primary Outcome: Response Rate During the First Course of JZP-458 Administration
Description: The response rate was defined as the number (proportion) of patients with the last 72-hour nadir serum asparaginase activity (NSAA) level ≥ 0.1 IU/mL during the first course of IM JZP-458. Blood samples were collected for serum asparaginase activity level determination.
Time Frame: Baseline up to 2 weeks
Population: Response rates were assessed in the Efficacy Analysis Set in participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: JZP-458 IM 25 mg/m^2 (MWF) | Part A: JZP-458 IM 37.5 mg/m^2 (MWF) | Part A: JZP-458 IM 25 (MW)/50 mg/m^2 (F) | Part B: JZP-458 IV 25 (MW)/50 mg/m^2 (F)
Number analyzed (Participants) | 28 | 77 | 49 | 50
Participants | 18 | 70 | 44 | 20

2. Primary Outcome: Number of Participants With Any Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered related to study drug. AEs were classified by the Investigator using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.
Time Frame: Date of written informed consent up to 30 days after last dose of last course, up to approximately 2 years 7 months
Population: Safety events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: JZP-458 IM 25 mg/m^2 (MWF) | Part A: JZP-458 IM 37.5 mg/m^2 (MWF) | Part A: JZP-458 IM 25 (MW)/50 mg/m^2 (F) | Part B: JZP-458 IV 25 (MW)/50 mg/m^2 (F)
Number analyzed (Participants) | 33 | 83 | 51 | 61
Participants | 32 | 83 | 49 | 60

3. Secondary Outcome: Number of Participants With Last 48-hour NSAA Level ≥ 0.1 IU/mL During The First Course (6 Doses) of JZP-458 Administration
Description: Blood samples were collected for serum asparaginase activity level determination.
Time Frame: Baseline up to 2 weeks
Population: Nadir serum asparaginase activity levels were assessed in the Efficacy Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: JZP-458 IM 25 mg/m^2 (MWF) | Part A: JZP-458 IM 37.5 mg/m^2 (MWF) | Part A: JZP-458 IM 25 (MW)/50 mg/m^2 (F) | Part B: JZP-458 IV 25 (MW)/50 mg/m^2 (F)
Number analyzed (Participants) | 32 | 83 | 49 | 59
Participants | 31 | 82 | 47 | 53

4. Secondary Outcome: Number of Participants With Last NSAA Levels ≥ 0.4 IU/mL During The First Course (6 Doses) of JZP-458 Administration
Description: Blood samples were collected for serum asparaginase activity level determination.
Time Frame: Baseline up to 2 weeks
Population: Nadir serum asparaginase activity levels were assessed in the Efficacy Analysis Set in participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: JZP-458 IM 25 mg/m^2 (MWF) | Part A: JZP-458 IM 37.5 mg/m^2 (MWF) | Part A: JZP-458 IM 25 (MW)/50 mg/m^2 (F) | Part B: JZP-458 IV 25 (MW)/50 mg/m^2 (F)
Number analyzed (Participants) | 32 | 83 | 49 | 59
Participants
  Last 48 hours | 16 | 65 | 32 | 10
  Last 72 hours: number analyzed (Participants) | 28 | 77 | 49 | 50
  Last 72 hours | 1 | 20 | 23 | 0

5. Secondary Outcome: Mean Serum Asparaginase Activity Levels in First Course of JZP-458 Administration
Description: Serum asparaginase levels serve as a surrogate marker for asparagine depletion. Mean serum asparaginase activity levels in Course 1 are reported.
Time Frame: Up to 2 weeks (6 doses)
Population: Serum asparaginase activity levels were assessed in participants with available data in the Efficacy Analysis Set.
Measure: Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Part A: JZP-458 IM 25 mg/m^2 (MWF) | Part A: JZP-458 IM 37.5 mg/m^2 (MWF) | Part A: JZP-458 IM 25 (MW)/50 mg/m^2 (F) | Part B: JZP-458 IV 25 (MW)/50 mg/m^2 (F)
Number analyzed (Participants) | 32 | 83 | 49 | 59
IU/mL
  Last 48 hours | 0.45 [0.37 to 0.53] | 0.88 [0.76 to 1.01] | 0.66 [0.54 to 0.77] | 0.25 [0.20 to 0.29]
  Last 72 hours: number analyzed (Participants) | 28 | 77 | 49 | 50
  Last 72 hours | 0.16 [0.12 to 0.19] | 0.33 [0.28 to 0.39] | 0.47 [0.35 to 0.59] | 0.10 [0.07 to 0.13]

6. Secondary Outcome: Number of Participants Who Are Anti-drug Antibody Positive or Negative Against JZP-458
Description: Blood samples were collected for immunogenicity analysis. Anti-drug antibody positive (ADA+) participants were those with a positive result on the first test and also a positive result on the confirmatory test. Anti-drug antibody negative (ADA-) participants had a negative result on the first test.
Time Frame: Baseline up to 30 days (ADA- samples) after last dose of last course and up to 6 months (ADA+ samples) after last dose of last course, up to approximately 2 years 7 months
Population: Immunogenicity was assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: JZP-458 IM 25 mg/m^2 (MWF) | Part A: JZP-458 IM 37.5 mg/m^2 (MWF) | Part A: JZP-458 IM 25 (MW)/50 mg/m^2 (F) | Part B: JZP-458 IV 25 (MW)/50 mg/m^2 (F)
Number analyzed (Participants) | 33 | 83 | 51 | 61
Participants
  Overall confirmed ADA+ | 16 | 41 | 25 | 34
  Overall ADA- | 17 | 42 | 26 | 27

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from date of written informed consent up to 30 days after last dose of last course, up to approximately 2 years 7 months.
Description: A treatment-emergent adverse event (TEAE) is defined as any event with onset date on or after the first dose of study treatment through the end of the study or any ongoing event that worsens in severity after the date of the first dose of study treatment through the end of the study.
Arm/Group | Part A: JZP-458 IM 25 mg/m^2 (MWF) | Part A: JZP-458 IM 37.5 mg/m^2 (MWF) | Part A: JZP-458 IM 25 (MW)/50 mg/m^2 (F) | Part B: JZP-458 IV 25 (MW)/50 mg/m^2 (F)
All-Cause Mortality (participants affected / at risk) | 1/33 | 2/83 | 0/51 | 0/61
Serious Adverse Events (participants affected / at risk) | 20/33 | 57/83 | 34/51 | 40/61
Other Adverse Events (participants affected / at risk) | 31/33 | 81/83 | 48/51 | 56/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: JZP-458 IM 25 mg/m^2 (MWF) (N=33) | Part A: JZP-458 IM 37.5 mg/m^2 (MWF) (N=83) | Part A: JZP-458 IM 25 (MW)/50 mg/m^2 (F) (N=51) | Part B: JZP-458 IV 25 (MW)/50 mg/m^2 (F) (N=61)
Febrile neutropenia (Blood and lymphatic system disorders) | 9 | 24 | 20 | 14
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Methaemoglobinaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 2 | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 1 | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 4 | 4 | 2
Vomiting (Gastrointestinal disorders) | 1 | 8 | 2 | 6
Nausea (Gastrointestinal disorders) | 2 | 6 | 1 | 4
Pancreatitis (Gastrointestinal disorders) | 0 | 3 | 3 | 2
Pancreatitis acute (Gastrointestinal disorders) | 0 | 4 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Anal inflammation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oesophageal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatic pseudocyst (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 3 | 8 | 8 | 3
Catheter site haemorrhage (General disorders) | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 1 | 0 | 0
Infusion site extravasation (General disorders) | 0 | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 2 | 4 | 2 | 5
Anaphylactic reaction (Immune system disorders) | 0 | 3 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 2 | 5 | 6 | 3
Enterocolitis infectious (Infections and infestations) | 0 | 2 | 3 | 0
Corona virus infection (Infections and infestations) | 2 | 0 | 2 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 2 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 2 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0
Skin infection (Infections and infestations) | 1 | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 1 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Anorectal infection (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 1
Citrobacter infection (Infections and infestations) | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0
Groin abscess (Infections and infestations) | 0 | 1 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0 | 0
Necrotising fasciitis (Infections and infestations) | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 1 | 3 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Anaphylactic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 1 | 1 | 2
Weight decreased (Investigations) | 0 | 0 | 2 | 1
Amylase increased (Investigations) | 0 | 0 | 1 | 0
Blood creatine increase (Investigations) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 1
Lipase increased (Investigations) | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0
Shigella test positive (Investigations) | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2
Blood culture positive (Investigations) | 0 | 0 | 0 | 1
Drug clearance decreased (Investigations) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 7 | 5 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 5
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Histiocytic sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
T-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Neurotoxicity (Nervous system disorders) | 0 | 1 | 2 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 2 | 0
Encephalopathy (Nervous system disorders) | 0 | 2 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1 | 1 | 0
Seizure (Nervous system disorders) | 0 | 2 | 0 | 2
Cerebrospinal fluid leakage (Nervous system disorders) | 1 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Leukoencephalopathy (Nervous system disorders) | 1 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Superior sagittal sinus thrombosis (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Hyperammonaemic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 1
Personality change (Psychiatric disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 4 | 3 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nephropathy toxic (Renal and urinary disorders) | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 2 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: JZP-458 IM 25 mg/m^2 (MWF) (N=33) | Part A: JZP-458 IM 37.5 mg/m^2 (MWF) (N=83) | Part A: JZP-458 IM 25 (MW)/50 mg/m^2 (F) (N=51) | Part B: JZP-458 IV 25 (MW)/50 mg/m^2 (F) (N=61)
Anaemia (Blood and lymphatic system disorders) | 13 | 47 | 28 | 22
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 5 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 4 | 0
Sinus bradycardia (Cardiac disorders) | 2 | 0 | 2 | 1
Sinus tachycardia (Cardiac disorders) | 5 | 17 | 7 | 4
Periorbital oedema (Eye disorders) | 2 | 1 | 0 | 0
Vision blurred (Eye disorders) | 2 | 3 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 5 | 25 | 13 | 9
Abdominal pain upper (Gastrointestinal disorders) | 3 | 3 | 2 | 3
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 3 | 0
Constipation (Gastrointestinal disorders) | 4 | 13 | 8 | 12
Diarrhoea (Gastrointestinal disorders) | 4 | 23 | 12 | 11
Dyspepsia (Gastrointestinal disorders) | 1 | 6 | 2 | 4
Gastrooesophageal reflux (Gastrointestinal disorders) | 4 | 1 | 3 | 3
Nausea (Gastrointestinal disorders) | 8 | 28 | 17 | 28
Oral pain (Gastrointestinal disorders) | 3 | 2 | 1 | 2
Pancreatitis (Gastrointestinal disorders) | 0 | 2 | 3 | 2
Stomatitis (Gastrointestinal disorders) | 6 | 22 | 14 | 17
Toothache (Gastrointestinal disorders) | 2 | 1 | 1 | 2
Vomiting (Gastrointestinal disorders) | 12 | 39 | 15 | 38
Asthenia (General disorders) | 2 | 1 | 1 | 0
Catheter site pain (General disorders) | 0 | 4 | 5 | 1
Catheter site rash (General disorders) | 0 | 2 | 0 | 4
Chills (General disorders) | 1 | 6 | 2 | 1
Fatigue (General disorders) | 10 | 32 | 13 | 15
Injection site pain (General disorders) | 3 | 4 | 3 | 0
Injection site reaction (General disorders) | 0 | 2 | 4 | 0
Pain (General disorders) | 4 | 6 | 0 | 2
Pyrexia (General disorders) | 8 | 31 | 11 | 12
Drug hypersensitivity (Immune system disorders) | 2 | 4 | 0 | 9
Corona virus infection (Infections and infestations) | 2 | 5 | 1 | 3
Enterocolitis infectious (Infections and infestations) | 2 | 1 | 1 | 1
Paronychia (Infections and infestations) | 2 | 0 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 7 | 2 | 9
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 6 | 4 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 2 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 4 | 8 | 8 | 3
Activated partial thromboplastin time prolonged (Investigations) | 1 | 7 | 3 | 1
Alanine aminotransferase increased (Investigations) | 6 | 29 | 10 | 18
Antithrombin III decreased (Investigations) | 0 | 1 | 3 | 0
Aspartate aminotransferase increased (Investigations) | 5 | 24 | 6 | 13
Blood alkaline phosphatase increased (Investigations) | 1 | 5 | 1 | 1
Blood bilirubin increased (Investigations) | 2 | 12 | 4 | 5
Blood cholesterol increased (Investigations) | 4 | 3 | 1 | 2
Blood creatinine increased (Investigations) | 0 | 8 | 3 | 5
Blood fibrinogen decreased (Investigations) | 3 | 3 | 0 | 1
CD4 lymphocytes decreased (Investigations) | 2 | 1 | 0 | 0
Haematocrit decreased (Investigations) | 2 | 1 | 2 | 0
Haemoglobin decreased (Investigations) | 2 | 1 | 0 | 1
Lymphocyte count decreased (Investigations) | 8 | 21 | 9 | 8
Neutrophil count decreased (Investigations) | 14 | 34 | 25 | 11
Platelet count decreased (Investigations) | 13 | 36 | 25 | 13
Weight decreased (Investigations) | 1 | 13 | 9 | 5
Weight increased (Investigations) | 2 | 1 | 0 | 3
White blood cell count decreased (Investigations) | 12 | 25 | 12 | 11
Decreased appetite (Metabolism and nutrition disorders) | 7 | 28 | 15 | 15
Dehydration (Metabolism and nutrition disorders) | 3 | 9 | 3 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 14 | 7 | 9
Hypermagnesemia (Metabolism and nutrition disorders) | 2 | 3 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 | 6 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 7 | 6 | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 12 | 3 | 6
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 9 | 4 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 6 | 1 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 14 | 11 | 8
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 5 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 7 | 4 | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 5 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 9 | 4 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 22 | 7 | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 7 | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 18 | 9 | 4
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1 | 1
Dizziness (Nervous system disorders) | 2 | 4 | 4 | 6
Headache (Nervous system disorders) | 12 | 23 | 12 | 11
Neuropathy peripheral (Nervous system disorders) | 1 | 5 | 2 | 2
Paraesthesia (Nervous system disorders) | 3 | 1 | 4 | 4
Peripheral motor neuropathy (Nervous system disorders) | 2 | 5 | 3 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 3 | 1 | 0
Tremor (Nervous system disorders) | 0 | 5 | 3 | 3
Agitation (Psychiatric disorders) | 3 | 4 | 1 | 2
Anxiety (Psychiatric disorders) | 2 | 9 | 5 | 7
Depression (Psychiatric disorders) | 1 | 5 | 2 | 0
Insomnia (Psychiatric disorders) | 5 | 8 | 3 | 8
Irritability (Psychiatric disorders) | 3 | 8 | 2 | 4
Mood swings (Psychiatric disorders) | 2 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 5 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 11 | 9 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 7 | 4 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 9 | 4 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 10 | 6 | 9
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 10 | 4 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 4 | 2 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1 | 4 | 3
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 | 6 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 6 | 3 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 3 | 5 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 2
Pruritis (Skin and subcutaneous tissue disorders) | 2 | 6 | 3 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 5 | 3 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 8 | 3 | 6
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 0
Flushing (Vascular disorders) | 4 | 4 | 3 | 0
Hypertension (Vascular disorders) | 1 | 6 | 8 | 2
Hypotension (Vascular disorders) | 1 | 6 | 2 | 2

LIMITATIONS AND CAVEATS:
Participants in this study received JZP-458 as part of a multi-agent chemotherapeutic regimen.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-03): https://cdn.clinicaltrials.gov/large-docs/31/NCT04145531/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/31/NCT04145531/SAP_002.pdf